CLINICAL TRIAL: NCT00243542
Title: ACZ ACN 01. A Phase 4, Double-Blind, Multicenter, Randomized, Vehicle-Controlled, Cross-Over Study to Further Evaluate the Risk of Hematological Adverse Events in G6PD-Deficient Subjects With Acne Vulgaris Treated With ACZONE™ (Dapsone) Gel, 5%.
Brief Title: Phase IV Study to Gather More Information About the Safety of ACZONE Gel, 5% in Treating Subjects With Acne Who Have G6PD Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ACZ ACN 01
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Acne Vulgaris
Keywords: Acne, G6PD deficiency, Dapsone
MeSH Terms: conditions — Acne Vulgaris; Glucosephosphate Dehydrogenase Deficiency

INTERVENTIONS:
Drug: ACZONE Gel, 5%
Drug: Vehicle

SUMMARY:
The purpose of this study is to gather more information about the safety of ACZONE Gel, 5% in treating subjects with acne who have certain blood disorders.

ACZONE Gel, 5% is a prescription skin use (topical) medicine used to help treat acne in people 12 years and older. ACZONE Gel, 5% has been studied in approximately 4000 people and was shown to reduce the number of pimples and improve acne.

The active drug ingredient in ACZONE Gel, 5% is dapsone. People with blood disorders called "G6PD deficiency", "methemoglobin reductase deficiency", and "hemoglobin M" have a higher chance of side effects with dapsone.

G6PD is short for "glucose-6-phosphate dehydrogenase". It is an enzyme found in red blood cells, which carry oxygen to all parts of the body. G6PD helps the red blood cells to function normally. Some people have less G6PD in their red blood cells than the average person. This is called G6PD deficiency.

Two treatments - ACZONE Gel, 5% and placebo - will be studied for comparison.

DETAILED DESCRIPTION:
Study Objectives:

* To compare the safety profile and risk of hemolysis of ACZONE Gel, 5% to that of the vehicle after 12 weeks each of twice daily applications in acne vulgaris subjects with glucose-6-phosphate-dehydrogenase (G6PD) deficiency.
* To determine the systemic levels of plasma dapsone and N-acetyl dapsone during treatment with ACZONE Gel, 5%.

Study Population:

Approximately 60 male and female subjects

Study Treatment:

All subjects in the study will receive ACZONE Gel, 5% and vehicle in 1 of 2 sequences; each for a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, subjects must fulfill all of the following criteria:

1. Male or female ≥12 years of age.
2. A clear diagnosis of acne vulgaris, defined as ≥20 acne inflammatory and/or non-inflammatory lesions (≥10 of the acne lesions must be on the face, the others may be present on the neck, shoulders, upper chest, and upper back) at screening.
3. A diagnosis of G6PD deficiency, defined as having a G6PD value below the lower limit of normal for the central reference laboratory.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. A dermal examination reveals the presence of severe cystic acne or acne conglobata.
2. Treatment with isotretinoin (Accutane®) within 3 months of baseline and throughout the study.
3. Subjects predisposed to anemia for other medical reasons, including but not limited to gastrointestinal bleeding and cancer.
4. Subjects who are using topical or systemic medications for acne throughout the study. This includes, but is not limited to, benzoyl peroxide, antibiotics, topical Vitamin A derivatives such as Retin-A.
5. Subjects who are using medication or eating foods that could potentially cause a hemolytic event in individuals with G6PD deficiency during the study.
6. Facial surgery (dermabrasion, laser resurfacing or other facial cosmetic surgeries) within 3 months of baseline and throughout the study.
7. A history of hypersensitivity to dapsone, parabens, or any component of the study products.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The within-subject between treatment period differences in change from baseline to the 2nd week of each treatment period and change from baseline to the end of each treatment period will be summarized based upon various lab parameters.
The safety evaluable data set will be used, and each variable will be summarized using descriptive statistics.
Analyses of clinical lab values, AEs, vitals, and concomitant meds will be performed on all subjects who received treatment.

SECONDARY OUTCOMES:
Acne Lesions: Tabular summaries of total lesion counts will be provided by appropriate descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Garrett, MS, DDS, Study Director — QLT USA, Inc.
Locations (29):
- United States (29):
  - Radiant Research, Inc., Birmingham, Alabama
  - Therapeutics Clinical Research, San Diego, California
  - Department of Dermatology, University of California, San Francisco, San Francisco, California
  - Dermatology Associates, PC at the Washington Hospital Center, Washington D.C., District of Columbia
  - Howard University Hospital Department of Dermatology, Washington D.C., District of Columbia
  - FXM Research, Miami, Florida
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Boston Clinical Trials, Boston, Massachusetts
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Washington University Dermatology Clinical Trials Unit, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Department of Dermatology SUNY Downstate Medical Center, Brooklyn, New York
  - Columbia University Medical Center Department of Dermatology, New York, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Universtiy Dermatology Consultants, Inc., Cincinnati, Ohio
  - Paddington Testing Clinic, Philadelphia, Pennsylvania
  - Society Hill Dermatology, Philadelphia, Pennsylvania
  - Okatie Research Center, LLC, Beaufort, South Carolina
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Dermatology Research Associates, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - DiscoveResearch, Inc., Beaumont, Texas
  - J&S Studies, Inc., Bryan, Texas
  - Research Across America, Dallas, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - The Education and Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Norfolk, Virginia
  - Advanced Healthcare, SC, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Piette WW, Taylor S, Pariser D, Jarratt M, Sheth P, Wilson D. Hematologic safety of dapsone gel, 5%, for topical treatment of acne vulgaris. Arch Dermatol. 2008 Dec;144(12):1564-70. doi: 10.1001/archdermatol.2008.518. PMID 19075138